CLINICAL TRIAL: NCT01570062
Title: Subclinical Cardiovascular Health Benefits of Interventions to Reduce Exposure to Combustion-Derived Particulate Air Pollution
Brief Title: Cardiovascular Effects of Aerosols in Residences Study
Acronym: CLEAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Ryan Allen, Assistant Professor, Simon Fraser University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Allen,R-MOP111042
Record Dates: First submitted 2012-03-15; First posted 2012-04-04 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Endothelial Dysfunction; Systemic Inflammation
Keywords: Inflammation; Pathologic Processes
MeSH Terms: conditions — Inflammation; Pathologic Processes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indoor Air HEPA Filtration (Active Comparator): HEPA filters will be placed in participant's main living area and bedroom. Actual filtration will occur during only one of the two 7-day sampling periods.
  Interventions: Device: HEPA Filter
- HEPA Filtration Placebo (Placebo Comparator): For one of two 7-day sampling sessions, HEPA filters placed in participants' homes will be run without an actual filter in the housing unit.
  Interventions: Device: HEPA Filtration Placebo

INTERVENTIONS:
Device: HEPA Filter — Two HEPA filters will be placed in participant's homes (one in the bedroom and one in the main living area); each HEPA will run for 2 consecutive 7-day sampling sessions. During one of the 7-day sampling sessions, the HEPA filter will run without the internal filter in place (i.e., "placebo" filtration).
  Other Names: Living area HEPA: Honeywell, Model 50250; Bedroom HEPA: Honeywell, Model 18155
  Arms: Indoor Air HEPA Filtration
Device: HEPA Filtration Placebo — for one of the two 7-day sampling sessions, both HEPA filters placed in participants' homes will be run without the actual filter in the housing unit.
  Other Names: Living area HEPA: Honeywell, Model 50250; Bedroom HEPA: Honeywell, Model 18155
  Arms: HEPA Filtration Placebo

SUMMARY:
This study is focused on the effects of HEPA filtration to reduce exposures to combustion-derived air pollution (CDAP). Specifically, the study will evaluate the health benefits of HEPA filters and compare the cardiovascular toxicity of two major sources of CDAP, specifically traffic and residential wood combustion.

Specifically, the purpose of this study is to evaluate the ability of portable high efficiency particle air (HEPA) filters to reduce exposures to PM2.5 and air pollution indoors and to improve subclinical indicators of microvascular function and systemic inflammation among healthy adult participants.

The investigators hypothesize that HEPA filter use will help decrease indoor concentrations of CDAP thereby helping to mitigate the associated cardiovascular risks.

DETAILED DESCRIPTION:
To address knowledge gaps about health risks of specific pollution sources and to provide new evidence on the health benefits of air pollution interventions, the objectives of this study are: 1) quantify the relationship between low-level exposures to combustion-derived PM air pollution and subclinical indicators of cardiovascular disease risk; and 2) compare the relative impact of HEPA filtration for two major PM sources (traffic and residential wood combustion) on these indicators.

The use of HEPA filters may help to mitigate cardiovascular risks factors caused by combustion-derived air pollution (CDAP), (specifically woodstove and traffic emissions). We hypothesize that HEPA filter use and improved woodstove technology will help decrease indoor occurrences of CDAP. This project will help address knowledge gaps in CDAP-related health risks and benefits of interventions. Specific objectives include establishing a relationship between exposure to CDAP and biomarkers of cardiovascular risk and evaluating the impact of HEPA filter use towards improved indoor air quality and health indicators.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* non-smoking household
* lives within study boundaries and in areas of interest

Exclusion Criteria:

* COPD
* asthma
* diabetes
* heart disease
* hypertension
* arthritis
* gum disease
* occupationally exposed to traffic exposures &/or woodsmoke
* if female, pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Difference in reactive hyperemia measurement after HEPA filtration | after 1 week of filtration
  Participants endothelial function are tested after 1 week of HEPA filtration and after 1 week of non-HEPA filtration (placebo filtration).

SECONDARY OUTCOMES:
Difference in C-Reactive Protein after HEPA Filtration | after 1 week of filtration
  Participants CRP is measured after 1 week of HEPA filtration and after 1 week of non-HEPA filtration (placebo filtration).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Allen, PhD, Principal Investigator — Simon Fraser University, Canada
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

REFERENCES:
- [Background] Allen RW, Carlsten C, Karlen B, Leckie S, van Eeden S, Vedal S, Wong I, Brauer M. An air filter intervention study of endothelial function among healthy adults in a woodsmoke-impacted community. Am J Respir Crit Care Med. 2011 May 1;183(9):1222-30. doi: 10.1164/rccm.201010-1572OC. Epub 2011 Jan 21. PMID 21257787
- [Derived] Kajbafzadeh M, Brauer M, Karlen B, Carlsten C, van Eeden S, Allen RW. The impacts of traffic-related and woodsmoke particulate matter on measures of cardiovascular health: a HEPA filter intervention study. Occup Environ Med. 2015 Jun;72(6):394-400. doi: 10.1136/oemed-2014-102696. Epub 2015 Apr 20. PMID 25896330